CLINICAL TRIAL: NCT03634696
Title: m-Palliative Care Link: Improving Symptom Control and Information Exchange Among Specialists and Local Health Workers Treating Late Stage Tanzanian Cancer Patients
Brief Title: m-Palliative Care Link: Improving Palliative Care for Late Stage Tanzanian Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susan Miesfeldt (Other)
Collaborators: MaineHealth (Other); National Institutes of Health (NIH) (NIH); Dimagi Inc. (Industry); Muhimbili University of Health and Allied Sciences (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor-Investigator, Susan Miesfeldt, Principal Investigator, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1040841; R21TW010190 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-08-16 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Cancer
Keywords: Late-stage; Palliative care; Novel technology; Communication
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Field test participants (Experimental): Late-stage adult cancer patients seeking care at Ocean Road Cancer Center, consenting to participate in mPCL application field test
  Interventions: Other: mPCL
- Control participants (Active Comparator): Late-stage adult cancer patients seeking care at Ocean Road Cancer Center, consenting to serve as controls for mPCL field test
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: mPCL — Smart phone application to support palliative care among late-stage cancer patients
  Arms: Field test participants
Other: Usual Care — Usual care through OCRI palliative care clinic
  Arms: Control participants

SUMMARY:
This work aims to improve late-stage cancer patients' access to high quality, patient-centered symptom assessment and control via the creation, field test, and outcomes assessment of a scalable mobile application (mPalliative Care Link; mPCL)-built around a locally-validated Palliative care Outcome Scale- that links a limited pool of existing Tanzanian palliative care specialists with patients, lay/family caregivers, and local health workers.

DETAILED DESCRIPTION:
The investigators hypothesize that a mobile device-based symptom assessment, control and communication application (m-Palliative Care Link (mPCL) will extend access to palliative care specialists (hereafter named specialists), resulting in: a) symptom control information exchange between specialists, patients, and local health workers and b) reduced symptom burden in late-stage cancer patients.

This hypothesis will be tested by accomplishing the following specific aims in the two-year study period:

Aim 1. In partnership with local palliative care specialists, to design and create a secure mobile communication application (m-Palliative Care Link; mPCL) for facilitating remote assessment of and communication about patient symptom control needs among specialists, patients/caregivers, and local health workers (all of whom are referred to here as user groups). mPCL will:

* Regularly deliver the APCA POS (hereafter POS) to the cancer patient/caregiver via mobile device; allow them to complete the outcome scale on this device; and return responses to the specialist and local health worker for access via a secure website.
* Enable specialist POS review/action in partnership with the local health worker.
* Allow the specialist to communicate with the patient/caregiver and local health worker regarding further symptom assessment and control based on existing standards and the patient's desires and needs.
* Enable the specialist to generate/update patient records for ongoing review.
* Record and track symptom control as a trajectory throughout the patient's illness via collection, storage, and analysis of POS responses.

Aim 2. To usability test an mPCL prototype through a combination of hands-on observation/feedback and survey-based assessment of ease of use and suggestions for change among 5-7 participants from each user group. Usability test data will be used to improve mPCL design for subsequent field test (see Aim 3).

Aim 3. To field test and validate usability of mPCL among 45 late-stage cancer patients. Late-stage cancer patients, who are eligible for the study, will be enrolled/consented, trained on mPCL use, and provided with an mPCL-equipped mobile device prior to discharge from ORCI. An mPCL record and discharge care plan will be generated by the specialist on his/her personal computer and communicated with the patient's local health worker for review and ongoing remote care communication and coordination. Field tests will continue for 4 months or until patient death. Through a combination of surveys and interviews of user groups, investigators will: determine the feasibility, acceptability, barriers, and facilitators of mPCL for communication and action regarding symptom assessment, information exchange, and symptom control; further optimize mPCL for ongoing study; determine the projected per patient cost of mPCL implementation; and gather rich data on the symptom control needs of Tanzanian cancer patients.

Aim 4. To collect preliminary data comparing field test symptom outcomes with 45 usual care patients (ORCI palliative care clinic patients). Patients will be identified, enrolled and consented during their scheduled outpatient clinic visit. POS responses will be collected at the time of each clinic visit for up to 4 months. Through examination/between-group comparisons (mPCL intervention versus usual care) of symptom-based outcomes and medication type, dose and duration, investigators will collect preliminary data on mPCL impact that is critical to design of a future large-scale, randomized mPCL outcomes study.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for field test if they meet the following criteria:

* Are ORCI inpatients with untreatable, late stage cancer
* Age 21 years or older
* Willing to enroll
* Able to understand and sign informed consent document
* Have four-month life expectancy or greater based on specialist assessment
* Have caregivers available/willing to support outpatient care for duration of field test
* Have a local health worker to support their outpatient care who consents to participate in the field test (i.e., partner with palliative care specialists for the duration of field test)
* Live within 50 km of ORCI for access to medications and study nurse support
* Have experience using a mobile device as measured by past cell phone ownership
* Have completed primary school

Exclusion Criteria:

• Not meeting inclusion criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Pain control | Up to 4 months
  APCA African Palliative Outcome Scale. Pain scale from 0-5 (low to high).

SECONDARY OUTCOMES:
Application utility | six week survey
  Survey delivered via smart phone to all application users.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Miesfeldt, MD, Principal Investigator — MaineHealth
Locations (1):
- Ocean Road Cancer Institute, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No